CLINICAL TRIAL: NCT03507569
Title: A Non-Randomized Open Label, Adaptive, Parallel Group, Human Positron Emission Tomography (PET) Study to Assess Occupancy of Brain alpha5-Containing GABAA Receptors of Ro7017773 Using [11C] Ro15-4513 Following Single Oral Doses in Healthy Participants
Brief Title: Open Label, Adaptive, Parallel Group PET Study Using RO7017773 And [11C] RO15-4513
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BP40257
Record Dates: First submitted 2018-04-16; First posted 2018-04-25 (Actual); Results first posted 2019-09-30 (Actual); Last update posted 2019-09-30 (Actual); Status verified 2019-08

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Ro 15-4513

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RO7017773 (Experimental): The first two participants of the first cohort are anticipated to receive a single dose of RO7017773 orally. The doses to be tested in the subsequent cohorts of participants will be determined by review of PET scan, PK, and safety results from the previous dose level.
  Interventions: Drug: RO7017773; Other: [11C] Ro15-4513

INTERVENTIONS:
Drug: RO7017773 — RO7017773 will be administered orally. The doses to be tested will be determined by review of PET scan, PK, and safety results from the previous dose level.
Other: [11C] Ro15-4513 — At the start of each PET scan, participants will receive an intravenous dose of the radiolabeled tracer [11C]Ro15-4513.

SUMMARY:
This is a single dose (SD), non-randomized, open-label, adaptive, parallel group study with the purpose of investigating the occupancy of alpha5-containing GABAA receptors by RO7017773 in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* Healthy (absence of evidence of any active or chronic disease following a detailed medical and surgical history, a complete physical examination including vital signs, 12-lead ECG, hematology, blood chemisty, serology, and urinalysis), as judged by the Investigator.
* Males and women of non-childbearing potential (WONCBP)

Exclusion Criteria:

* History of convulsions (other than benign febrile convulsions of childhood) including epilepsy, or personal history of significant cerebral trauma or CNS infections
* Clinically significant abnormal finding from the MRI performed after the initial screening examination
* Abnormal blood pressure, i.e, systolic blood pressure (SBP) greater than 140 or less than 90 mm Hg, and diastolic blood pressure (DBP) greater than 90 or less than 50 mm Hg
* Abnormal pulse rate, resting pulse rate greater than 100 or less than 40 bpm
* History or presence of clinically significant ECG abnormalities before study drug administration or cardiovascular disease
* Show evidence of human immunodeficiency virus (HIV) infection and/or positive human HIV antibodies
* Positive result on hepatitis B (HBV) or hepatitis C (HCV), presence of hepatitis B surface antigen (HBsAg) or positive hepatitis C antibody test result at screening or within 3 months prior to starting study treatment

Ages: 23 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2018-04-24 (Actual); Primary Completion 2018-06-22 (Actual); Study Completion 2018-06-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Hammersmith Medicines Research; Central Middlesex Hospital, London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy subjects between the ages of 23 and 55 years (inclusive) were enrolled at one site in the United Kingdom.
Groups:
- RO7017773 - 15mg; RO7017773 - 30mg; RO7017773 - 75mg; RO7017773 - 375mg: Healthy participants received a single oral dose of RO7017773, and up to 3 intravenous (IV) doses of the radiolabeled ligand [11C]Ro15-4513 administered prior to positron emission tomography/computed tomography (PET/CT) scans over two imaging sessions separated by at least 7 days.
Period: Overall Study
Arm/Group | RO7017773 - 15mg | RO7017773 - 30mg | RO7017773 - 75mg | RO7017773 - 375mg
Started | 2 | 1 | 2 | 1
Completed | 2 | 1 | 2 | 1
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | RO7017773 - 15mg | RO7017773 - 30mg | RO7017773 - 75mg | RO7017773 - 375mg | Total
Number analyzed (Participants) | 2 | 1 | 2 | 1 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: This data/information can potentially be used to re-identify trial participants due to the low sample size, Therefore, this data will not be disclosed in the interest of maintaining participant confidentiality.
Sex: Female, Male [Count of Participants; unit: Participants] — Population: This data/information can potentially be used to re-identify trial participants due to the low sample size, Therefore, this data will not be disclosed in the interest of maintaining participant confidentiality.
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: This data/information can potentially be used to re-identify trial participants due to the low sample size, Therefore, this data will not be disclosed in the interest of maintaining participant confidentiality.
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: This data/information can potentially be used to re-identify trial participants due to the low sample size, Therefore, this data will not be disclosed in the interest of maintaining participant confidentiality.

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Brain Alpha5-Containing GABA-A Receptors Occupied by RO7017773
Time Frame: Baseline up to 48 hours (hrs)
Population: This data/information can potentially be used to re-identify trial participants due to the low sample size, Therefore, this data will not be disclosed in the interest of maintaining participant confidentiality.
Arm/Group | RO7017773 - 15mg | RO7017773 - 30mg | RO7017773 - 75mg | RO7017773 - 375mg
Number analyzed (Participants) | 0 | 0 | 0 | 0

2. Primary Outcome: Plasma Concentrations of RO7017773
Time Frame: Baseline up to 48 hrs
Population: as for outcome 1
Arm/Group | RO7017773 - 15mg | RO7017773 - 30mg | RO7017773 - 75mg | RO7017773 - 375mg
Number analyzed (Participants) | 0 | 0 | 0 | 0

3. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Time Frame: From treatment initiation until 14 days after the last dose of study treatment.
Measure: Number; unit: Participants
Arm/Group | RO7017773 - 15mg | RO7017773 - 30mg | RO7017773 - 75mg | RO7017773 - 375mg
Number analyzed (Participants) | 2 | 1 | 2 | 1
Participants | 2 | 0 | 1 | 1

ADVERSE EVENTS:
Time Frame: From treatment initiation until 14 days after the last dose of study treatment.
Description: All participants randomized to study treatment and who received at least one dose of the study treatment, whether prematurely withdrawn from the study or not, were included in the safety analysis.
Arm/Group | RO7017773 - 15mg | RO7017773 - 30mg | RO7017773 - 75mg | RO7017773 - 375mg
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/1 | 0/2 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/1 | 0/2 | 0/1
Other Adverse Events (participants affected / at risk) | 2/2 | 0/1 | 1/2 | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RO7017773 - 15mg (N=2) | RO7017773 - 30mg (N=1) | RO7017773 - 75mg (N=2) | RO7017773 - 375mg (N=1)
Catheter site pain (General disorders) | 2 | 0 | 0 | 0
Catheter site paraesthesia (General disorders) | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Catheter site bruise (General disorders) | 0 | 0 | 0 | 1
Muscle contractions involuntary (Nervous system disorders) | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-08): https://cdn.clinicaltrials.gov/large-docs/69/NCT03507569/Prot_SAP_000.pdf